CLINICAL TRIAL: NCT01119300
Title: EUropean Pharmacogenetics of AntiCoagulant Therapy - Warfarin
Acronym: EU-PACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Collaborators: Utrecht University (Other); Leiden University Medical Center (Other); Erasmus Medical Center (Other); University of Ulm (Other); Newcastle University (Other); University of Liverpool (Other); LGC Limited (Industry); Uppsala University (Other); Democritus University of Thrace (Other); Elisabethinen Hospital (Other)
Responsible Party: Principal Investigator, Anke-Hilse Maitland-van der Zee, PharmD, PhD, Utrecht Institute for Pharmaceutical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: COU-001W
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Venous Thromboembolism; Atrial Fibrillation
Keywords: Venous Thromboembolism (VTE); Atrial Fibrillation (AF)
MeSH Terms: conditions — Venous Thromboembolism; Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Standard care
  Interventions: Other: Standard care
- Genotype-guided dosing algorithm (Experimental): Genotyping for CYP2C9*2, CYP2C9*3, and VKORC1 (-1639G→A) was performed with the use of a point-of-care test. For patients assigned to the genotype-guided group, warfarin doses were prescribed according to pharmacogenetic-based algorithms for the first 5 days.
  Interventions: Other: Genotype-guided dosing algorithm

INTERVENTIONS:
Other: Genotype-guided dosing algorithm — Loading and monitoring dose according to genotype-guided dosing algorithm
  Arms: Genotype-guided dosing algorithm
Other: Standard care — Standard care
  Arms: Standard care

SUMMARY:
Rationale:

The narrow therapeutic range and wide inter-patient variability in dose requirement make anticoagulation response to coumarin derivatives unpredictable. As a result, patients require frequent monitoring to avert adverse effects and maintain therapeutic efficacy. Polymorphisms in cytochrome P450 2C9 (CYP2C9) and vitamin K epoxide reductase complex 1 (VKORC1) jointly account for about 40% of the inter-individual variability in dose requirements. To date, several pharmacogenetic guided dosing algorithms for coumarin derivatives, predominately for warfarin, have been developed. However, the potential benefit of these dosing algorithms in terms of their safety and clinical utility has not been adequately investigated in randomised settings. Objective:

To determine whether a dosing algorithm containing genetic information increases the time within therapeutic INR range during anticoagulation therapy with each of warfarin, acenocoumarol and phenprocoumon compared to a dosing regimen that does not contain this information. Secondary outcomes of the study include cost effectiveness, number of thromboembolic and bleeding events, time to reach stable dose and number of supratherapeutic INR peaks.

DETAILED DESCRIPTION:
Study design: This is a two-armed, single-blinded, randomised controlled trial. In one arm (intervention) patients commencing anticoagulation therapy with either warfarin, acenocoumarol or phenprocoumon will be dosed according to a drug-specific genotype-guided dosing algorithm, which is based on genetic information, clinical data and (in the monitoring phase) previous INR. For the other arm (control) patients will be dosed according to a non-genotype-guided dosing regimen which does not include genetic information. The follow-up period per patient is 3 months. Study population: Newly diagnosed patients of both genders and at least 18 years old who need anticoagulant treatment with either acenocoumarol, phenprocoumon or warfarin within the low intensity INR range will be included in the trial. Main study parameters/endpoints: The % time within therapeutic INR range in the first 3 months of anticoagulation therapy. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Six extra blood samples are taken from each participant at the start of the study. Patients also have to attend 8 scheduled visits within the 3 months study period and are asked to fill in questionnaires. The genotype-guided dosing algorithm is anticipated to improve the accuracy of coumarin dosing and thus improve the safety and efficacy of anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either venous thromboembolism (VTE) or atrial fibrillation (AF) requiring coumarin therapy for at least 12 weeks and a target INR in the low intensity range (INR range 2-3 in the United Kingdom, Sweden, Germany, Austria and Greece and INR 2.5-3.5 in the Netherlands)
* Age ≥ 18 years
* Ability to attend scheduled visits
* Signed informed consent

Exclusion Criteria:

* Presence of a mechanical heart valve
* Severe cognitive impairment
* Known genotype CYP2C9 or VKORC1 at start of the study
* Previous or current treatment with any coumarin
* Pregnancy or lactation
* Non-eligible subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percent time within therapeutic INR range 2-3 during 12 weeks following the initiation of coumarin therapy | 12 weeks

SECONDARY OUTCOMES:
Time INR > or = 4.0, which indicates overanticoagulation | 12 weeks
Percent time spent > or = INR 4.0 | 12 weeks
Percent time spent < or = INR 2, which indicates under-anticoagulation | 12 weeks
Time to reach therapeutic INR defined as the time to the first INR within target range, providing that a subsequent INR > or =1 week later is also within target range | 12 weeks
Time to reach stable dose defined as INR within target range for a period of at least 3 weeks with <10% change in dose | 12 weeks
Time to and number of minor and major bleeding events | 12 weeks
Time to and number of thromboembolic events (therapeutic failure) | 12 weeks
The incidence of coumarin sensitivity | 12 weeks
The incidence of coumarin resistance | 12 weeks
Number of coumarin dose adjustments | 12 weeks
The clinical utility of the rapid genotyping test developed by LGC | 2 years
Quality of life as reported by the patient tested by the EuroQol (EQ)-5D questionnaire | 12 weeks
The cost-effectiveness of genotype-guided dosing for each coumarin compared with non-genotype-guided dosing | will be assessed after inclusion of all patients
Number of patients with INR > or = 4.0, which indicates overanticoagulation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Munir Pirmohamed, MD PhD, Principal Investigator — University of Liverpool
Locations (3):
- Uppsala University, Uppsala, Sweden
- United Kingdom (2):
  - University of Liverpool, Liverpool
  - University of Newcastle, Newcastle

REFERENCES:
- [Background] van Schie RM, Wadelius MI, Kamali F, Daly AK, Manolopoulos VG, de Boer A, Barallon R, Verhoef TI, Kirchheiner J, Haschke-Becher E, Briz M, Rosendaal FR, Redekop WK, Pirmohamed M, Maitland van der Zee AH. Genotype-guided dosing of coumarin derivatives: the European pharmacogenetics of anticoagulant therapy (EU-PACT) trial design. Pharmacogenomics. 2009 Oct;10(10):1687-95. doi: 10.2217/pgs.09.125. PMID 19842940
- [Background] Verhoef TI, Redekop WK, Darba J, Geitona M, Hughes DA, Siebert U, de Boer A, Maitland-van der Zee AH, Barallon R, Briz M, Daly A, Haschke-Becher E, Kamali F, Kirchheiner J, Manolopoulos VG, Pirmohamed M, Rosendaal FR, van Schie RM, Wadelius M; EU-PACT Group. A systematic review of cost-effectiveness analyses of pharmacogenetic-guided dosing in treatment with coumarin derivatives. Pharmacogenomics. 2010 Jul;11(7):989-1002. doi: 10.2217/pgs.10.74. PMID 20602617
- [Background] van Schie RM, Jorgensen AL, de Boer A, Maitland-van der Zee AH; EU-PACT study group. Systematic review of pharmacogenetic warfarin dosing. J Gen Intern Med. 2009 Oct;24(10):1171. doi: 10.1007/s11606-009-1083-9. No abstract available. PMID 19693633
- [Background] van Schie RM, Verhoef TI, Boejharat SB, Schalekamp T, Wessels JA, le Cessie S, Rosendaal FR, van der Meer FJ, de Boer A, Maitland-van der Zee AH. Evaluation of the effect of statin use on the acenocoumarol and phenprocoumon maintenance dose. Drug Metabol Drug Interact. 2012;27(4):229-34. doi: 10.1515/dmdi-2012-0024. PMID 23096528
- [Background] Verhoef TI, Redekop WK, Hegazy H, de Boer A, Maitland-van der Zee AH; EU-PACT group. Long-term anticoagulant effects of CYP2C9 and VKORC1 genotypes in phenprocoumon users. J Thromb Haemost. 2012 Dec;10(12):2610-2. doi: 10.1111/jth.12007. No abstract available. PMID 23016521
- [Background] Verhoef TI, Redekop WK, van Schie RM, Bayat S, Daly AK, Geitona M, Haschke-Becher E, Hughes DA, Kamali F, Levin LA, Manolopoulos VG, Pirmohamed M, Siebert U, Stingl JC, Wadelius M, de Boer A, Maitland-van der Zee AH; EU-PACT group. Cost-effectiveness of pharmacogenetics in anticoagulation: international differences in healthcare systems and costs. Pharmacogenomics. 2012 Sep;13(12):1405-17. doi: 10.2217/pgs.12.124. PMID 22966889
- [Background] van Schie RM, el Khedr N, Verhoef TI, Teichert M, Stricker BH, Hofman A, Buhre PN, Wessels JA, Schalekamp T, le Cessie S, van der Meer FJ, Rosendaal FR, de Boer A, Maitland-van der Zee AH, Visser LE. Validation of the acenocoumarol EU-PACT algorithms: similar performance in the Rotterdam Study cohort as in the original study. Pharmacogenomics. 2012 Aug;13(11):1239-45. doi: 10.2217/pgs.12.101. PMID 22920394
- [Background] van Schie RM, Babajeff AM, Schalekamp T, Wessels JA, le Cessie S, de Boer A, van der Meer FJ, van Meegen E, Verhoef TI, Rosendaal FR, Maitland-van der Zee AH; EU-PACT study group. An evaluation of gene-gene interaction between the CYP2C9 and VKORC1 genotypes affecting the anticoagulant effect of phenprocoumon and acenocoumarol. J Thromb Haemost. 2012 May;10(5):767-72. doi: 10.1111/j.1538-7836.2012.04694.x. PMID 22409277
- [Background] Verhoef TI, Redekop WK, Buikema MM, Schalekamp T, Van Der Meer FJ, Le Cessie S, Wessels JA, Van Schie RM, De Boer A, Teichert M, Visser LE, Maitland-Van Der Zee AH; EU-PACT Group. Long-term anticoagulant effects of the CYP2C9 and VKORC1 genotypes in acenocoumarol users. J Thromb Haemost. 2012 Apr;10(4):606-14. doi: 10.1111/j.1538-7836.2012.04633.x. PMID 22252093
- [Background] Avery PJ, Jorgensen A, Hamberg AK, Wadelius M, Pirmohamed M, Kamali F; EU-PACT Study Group. A proposal for an individualized pharmacogenetics-based warfarin initiation dose regimen for patients commencing anticoagulation therapy. Clin Pharmacol Ther. 2011 Nov;90(5):701-6. doi: 10.1038/clpt.2011.186. Epub 2011 Sep 28. PMID 22012312
- [Background] van Schie RM, Wessels JA, le Cessie S, de Boer A, Schalekamp T, van der Meer FJ, Verhoef TI, van Meegen E, Rosendaal FR, Maitland-van der Zee AH; EU-PACT Study Group. Loading and maintenance dose algorithms for phenprocoumon and acenocoumarol using patient characteristics and pharmacogenetic data. Eur Heart J. 2011 Aug;32(15):1909-17. doi: 10.1093/eurheartj/ehr116. Epub 2011 Jun 2. PMID 21636598
- [Background] van Schie RM, Wessels JA, Verhoef TI, Schalekamp T, le Cessie S, van der Meer FJ, Rosendaal FR, Visser LE, Teichert M, Hofman A, Buhre PN, de Boer A, Maitland-van der Zee AH. Evaluation of the effect of genetic variations in GATA-4 on the phenprocoumon and acenocoumarol maintenance dose. Pharmacogenomics. 2012 Dec;13(16):1917-23. doi: 10.2217/pgs.12.174. PMID 23215884
- [Background] Verhoef TI, Zuurhout MJ, van Schie RM, Redekop WK, van der Meer FJ, le Cessie S, Schalekamp T, de Boer A, Maitland-van der Zee AH. The effect of omeprazole and esomeprazole on the maintenance dose of phenprocoumon. Br J Clin Pharmacol. 2012 Dec;74(6):1068-9. doi: 10.1111/j.1365-2125.2012.04295.x. No abstract available. PMID 22497277
- [Background] van Schie RM, de Boer A, Maitland-van der Zee AH. Implementation of pharmacogenetics in clinical practice is challenging. Pharmacogenomics. 2011 Sep;12(9):1231-3. doi: 10.2217/pgs.11.81. No abstract available. PMID 21919599
- [Background] van Schie RM, Cascorbi I, Maitland-van der Zee AH. Conference Scene: Pharmacogenomics at the second PharmSciFair 2009: adverse drug reactions and clinical implementation. Pharmacogenomics. 2009 Sep;10(9):1389-91. doi: 10.2217/pgs.09.95. PMID 19761363
- [Result] Pirmohamed M, Burnside G, Eriksson N, Jorgensen AL, Toh CH, Nicholson T, Kesteven P, Christersson C, Wahlstrom B, Stafberg C, Zhang JE, Leathart JB, Kohnke H, Maitland-van der Zee AH, Williamson PR, Daly AK, Avery P, Kamali F, Wadelius M; EU-PACT Group. A randomized trial of genotype-guided dosing of warfarin. N Engl J Med. 2013 Dec 12;369(24):2294-303. doi: 10.1056/NEJMoa1311386. Epub 2013 Nov 19. PMID 24251363